





Asthma: Phenotyping Exacerbations 3

10TH November 2021







## **CONSENT FORM** (Final version 1.0: 10.11.2021)

Title of Study: Asthma: Phenotyping Exacerbations 3

IRAS Project ID: 304615

Name of Researcher: Dr Matthew Martin

| Name of Participant: Please | | | | e <u>initial</u> box |
|---|---|---|---|---|
| 1. | I confirm that I have read and undidated 10.11.2021 for the above s | | | 0 |
| 2. | I understand that my participation without giving any reason, and w understand that should I withdraw and that this information may still | vithout my medical car | e or legal rights being affected. collected so far cannot be erase | , 🗀 |
| 3. | I understand that relevant sections of my medical notes and data collected in the study may be looked at by authorised individuals from the University of Nottingham, the research group and regulatory authorities where it is relevant to my taking part in this study. I give permission for these individuals to have access to these records and to collect, store, analyse and publish information obtained from my participation in this study. I understand that my personal details will be kept confidential. | | | |
| 4. | I understand and agree that nasal brush samples will be taken for DNA and RNA extraction and genetic analysis (Optional) | | | |
| 5. | Consent for storage and use in possible future research (Optional) I agree that the samples I have given and the information gathered about me can be stored by the University of Nottingham at the Division of Respiratory Medicine, for possible use in future studies. I understand that some of these studies may be carried out by researchers other than the current team who ran the first study, including researchers working for commercial companies. Any samples or data used will be anonymised, and I will not be identified in anyway. | | | |
| 6. | 6. I agree to my GP being informed of my participation in this study and of any incidental findings. | | | |
| 7. | 7. I agree to take part in the above study. | | | |
| Na | ame of Participant | Date | Signature | |
| Na | ame of Person taking consent | Date | Signature | |

4 copies: 1 for participant, 1 for the project notes, 1 for the medical notes and 1 for HTA.